CLINICAL TRIAL: NCT01008787
Title: Peer-support Motivational Interviewing Physical Activity Intervention for African American Women
Brief Title: Motivational Interviewing for Physical Activity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-0257; NCI-2012-02123 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer Prevention; Focus Group; Interview; Physical Activity; African American women; Exercise; Exercise habits; Health behavior
MeSH Terms: conditions — Neoplasms; Motor Activity; Health Behavior | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- Focus Group (No Intervention): Qualitative interviews examining social support for PA conducted with African American (AA) women recruited from Wheeler Avenue Baptist Church located in Houston used to design Culturally-Appropriate Peer-based Motivational Interviewing (CAPMI) intervention.
- Intervention Group 1 (Active Comparator): CAPMI Intervention: Training + Weekly Partner Questionnaire + Interview + PA Newsletter
  Interventions: Behavioral: Training; Behavioral: Questionnaire; Behavioral: Interview; Behavioral: PA Newsletter
- Intervention Group 2 (Active Comparator): Interview + PA Newsletter
  Interventions: Behavioral: Interview; Behavioral: PA Newsletter

INTERVENTIONS:
Behavioral: Training — In-person 8-hour group physical activity training session (either over 1 or 2 days) and receive workbook and pedometer.
  Arms: Intervention Group 1
Behavioral: Questionnaire — Weekly during Weeks 2-7, complete question form given at training course about conversations with study partner, 5 minutes to complete.
  Arms: Intervention Group 1
Behavioral: Interview — Weeks 4 and 8, 30 minute phone interview about mood and physical activity.
  Arms: Intervention Group 1; Intervention Group 2
Behavioral: PA Newsletter — At Weeks 5 and 9, receive a physical activity (PA) newsletter.
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
The goal of this behavioral research study is to learn why some African American (AA) women choose not to exercise often and to learn if teaching African American women how to support the exercise habits of a partner will increase their physical activity and help them to stay more active over time.

The primary goal of the proposed intervention is:

Aim 1: To conduct formative research using semi-structured in-depth interviews and focus groups with sedentary AA women to investigate the role and importance of social support for PA;

Aim 2: To determine the feasibility of recruiting and implementing "Culturally Appropriate Physical Activity Motivational Interviewing" (CAPMI) intervention in sedentary AA women;

Aim 3: To pilot test and evaluate the efficacy of the CAPMI in increasing PA, social support, self-efficacy and reducing barriers to Physical Activity (PA) at post-intervention compared to an attention control group.

DETAILED DESCRIPTION:
Focus Group:

If you agree to take part in this study, you will take part in a focus group or individual interview. A focus group is a group of people who are asked questions about certain topics and then discuss these topics with other group members. During the focus group, you will talk about ways that African American women may increase their physical activity. You will also be asked questions about the ways in which you support other women to help them become more physically active. There will be 4 focus groups, each made up of 8-10 women. The focus group session should take 1 1/2 to 2 hours.

The focus group will be audiotaped and transcribed (the spoken words will be typed up). Your individual name will not be used during the focus group and will not be recorded. For example, you will be listed as Participant #1. After the focus group comments are copied down, the focus group tapes will be destroyed. The study staff may also interview you alone. During the individual interview, you will talk about ways that African American women may increase their physical activity. You will also be asked questions about the ways in which you support other women to help them become more physically active. The staff will interview 10 women. The individual interview should take 1 1/2 to 2 hours.

The individual interview will be audiotaped and transcribed. Your individual name will not be used during the interview and will not be recorded. For example, you will be listed as Participant #1. After the interview comments are copied down, the interview tapes will be destroyed.

Length of Study:

You will be on study until you complete the focus group session.

This is an investigational study. Up to 40 women will take part in the focus groups. All will be enrolled at M. D. Anderson.

Intervention:

You will need a partner (a female friend or family member) to take part in this study. Both you and your study partner will need to meet the same eligibility requirements, and both of you will be enrolled as participants. If you choose a partner that is not eligible, you will will need to choose another eligible partner before you can be enrolled in the study.

Screening:

Before you can take part in this study, you will be asked if you are between the ages of 18 and 65 years old, if you are currently not engaging in physical activity for more than 3 days per week and more than 20 minutes each day, and if you are ready to be physically active. You will be asked if you have a home address where information can be mailed, are able to read at a 6th grade level, and are able to participate in a training course that will take place on a weekend.

You will also be asked if you are pregnant or plan to become pregnant during the next 12 weeks. You will also be asked if you plan to move outside of the Houston area in the next 12 weeks. If you are pregnant, plan to become pregnant, and/or plan to move, you will not be able to take part in this study.

Baseline Tests:

If you are found to be eligible to take part in this study, you will complete the following tests and procedures:

* You will be asked how you are feeling and how often you exercise.
* Your height and weight will be measured.
* You will fill out a questionnaire about issues related to your physical activity. It will take 45-60 minutes to complete.
* You will take a walking test, in which you will walk for 6 minutes at a comfortable pace.
* You will receive a pedometer (a monitor that shows how far you walk).
* You may receive an accelerometer and complete a 7-day accelerometer assessment. An accelerometer is a small device that is worn on your hip that measures the amount of physical activity you do.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to either group.

Group 1:

If you are in Group 1, you will take part in an 8-hour training course conducted as 2 in-person 4-hour sessions (for example, scheduled on 2 Saturdays in a row) to help you learn how to support the exercise habits of your study partner. At this course, a trainer will give you information and you will take part in activities with your study partner. Sample activities include role playing and watching a video. This will take place on a weekend. The goal of the training course is to help you and your partner engage in physical activity. You will be asked to be physically active for 30 minutes each day.

You will receive a workbook and a DVD about physical activity. You will also be given a form to complete each time you speak with your study partner about physical activity. You will be asked to speak with your partner at least 1 time a week about your physical activities.

Each week during Weeks 1-4, 8, and 12 you will be asked to answer questions on the form given to you at the training course about the conversations you have with your study partner, and to complete recorded conversations via toll-free number. All telephone diaries must be completed and returned to research staff members by week 12 of the study.

At Weeks 4 and 8, you will be called and asked several questions about your mood and your physical activity. The phone call should take about 45 minutes.

At Weeks 5 and 9, you will be mailed a physical activity newsletter.

Group 2:

If you are in Group 2, at Weeks 4 and 8, you will be called and asked several questions about your mood and your physical activity. The phone call should take about 45 minutes.

At Weeks 5 and 9, you will receive a physical activity newsletter.

End-of-Study Visit:

At Week 12 of the study, you will complete the following tests and procedures:

* You will be asked several questions about your mood and your physical activity.
* Your height and weight will be measured.
* You will take a walking test, in which you will walk for 6 minutes at a comfortable pace.
* You may receive an accelerometer and complete a 7-day accelerometer assessment. An accelerometer is a small device that is worn on your hip that measures the amount of physical activity you do.

Length of Study You will be on study for 12 weeks.

This is an investigational study. Up to 80 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. African American (AA) woman (self-defined by participant) ages 18-65 years
2. Currently sedentary, defined as self-reported PA <3 days/week for <20 minutes/day over the past 6 months
3. Be ready and physically able to start being physically active, i.e., in preparation stage of change.
4. Have a home address where information can be mailed and working telephone.
5. Able to read English at a sixth-grade level as assessed by the Rapid Estimate of Adult Literacy in Medicine (REALM)
6. Identify a sedentary AA female (i.e., non-intimate family member or friend) with whom they can enroll in the study
7. Both partners are required to meet the same eligibility requirements and both partners will be enrolled as participants. Each woman will complete the same consent form.
8. Be available to participate in weekend trainings

Exclusion Criteria:

1. Currently taking medication for blood pressure or heart condition, or other physical limitations that might be aggravated by participation in moderate-intensity PA as measured using the PA Readiness Questionnaire
2. Pregnant or thinking about becoming pregnant during the study period
3. Thinking about moving to a location outside the greater Houston area during the study period
4. Being unable to attend the CAPMI training sessions with their partner
5. Participated in Phase I focus group/interviews
6. Being a male

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported Minutes of Moderate-intensity Physical Activity per Week | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, PhD, MPH, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org